CLINICAL TRIAL: NCT05149469
Title: Evaluation of Preimplantation Genetic Diagnosis for Neurofibromatosis Type 1 (NF1), Emphasizing on the Molecular Aspects
Brief Title: Molecular Aspects of Preimplantation Genetic Diagnosis for NF1
Acronym: NF1
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8374
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis Type 1; NF1; Preimplantation genetic diagnosis; De novo mutation; Mosaicism; Molecular test
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurofibromatosis 1 (NF1) is a multisystem disorders characterized by skin abnormalities, such as café-au-lait spots and neurofibromas, learning disabilities, skeletal anomalies and vascular complications. Experience learns that this disorder is a great burden for patients. NF1 is an autosomal dominant disorder with 50% risk of transmission. The penetrance is nearly 100%, but the expression varies greatly even within families, which makes it nearly impossible to predict severity in offspring. Preimplantation genetic diagnosis (PGD) is a reproductive option for couples at risk of transmitting NF1 to their offspring. We perform a retrospective and observational multicentric study in the Maastricht University Medical Center, the University Hospital of Brussel and Strasbourg University Hospital. Our specific (and first) goal is to evaluate the molecular aspects of PGD for NF1 in an international cohort of couples requesting PGD for NF1.

About 50% of the patients with NF1 have a de novo mutation that can complicate development of a PGD test. Earlier studies from 1990 and 1992 have shown that de novo NF1 mutations usually occur on the paternal allele. We want to confirm these findings with collected data from our cohort. The high incidence of de novo mutations results in a higher chance of finding mosaicism in patients or their parents. As a result of this, it can become apparent during PGD test preparation that PGD treatment is no longer possible or indicated. The investigators will evaluate these aspects of PGD for NF1 in our cohort.

They are also interested, as a second goal, in other aspects of PGD treatment for NF1, such as the success rate in thier cohort. They expect the success rate to be the same as for other autosomal dominant disorders

ELIGIBILITY:
Inclusion criteria:

* Major subjects (≥18 years old)
* Couples who have been treated at the HUS for a preimplantation diagnosis request for type 1 neurofibromatosis (confirmed by a molecular molecular analysis) and who have benefited from preliminary analyzes, between 01/01/2004 and 30/06 / 2021
* Couple who, after receiving information, did not express their opposition to the reuse of their data for the purposes of this research

Exclusion criteria:

* Couples who expressed their opposition to participating in the study
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Major subjects (≥18 years old) who have been treated at the HUS for a preimplantation diagnosis request for type 1 neurofibromatosis (confirmed by a molecular molecular analysis) and who have benefited from preliminary analyzes, between 01/01/2004 and 30/06 / 2021
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Study of the molecular aspects of PGD for NF1 in a large European cohort. | Files analysed retrospectively from from January 1, 2004 to June 30, 2021 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service Laboratoire de Diagnostic Génétique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France